CLINICAL TRIAL: NCT06330558
Title: Side-specific Factors for Conversion in Adrenalectomy for Pheochromocytoma. A Comparative Analysis
Brief Title: Side-specific Factors for Conversion in Adrenalectomy for Pheochromocytoma.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: pheos
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Adrenal Tumor
MeSH Terms: conditions — Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: laparoscopic right adrenalectomy
  Interventions: Procedure: laparoscopic right adrenalectomy
- Group B: laparoscopic left adrenalectomy
  Interventions: Procedure: laparoscopic right adrenalectomy

INTERVENTIONS:
Procedure: laparoscopic right adrenalectomy — adrenalectomy

SUMMARY:
Context: Adrenalectomy for pheochromocytoma (PHEO) poses difficulties due to the elevated chance of conversion. The objective of this study was to conduct a comparative analysis of the occurrence and determinants of conversion in left-sided abdominal laparoscopic adrenalectomy (LLA) and right-sided abdominal laparoscopic adrenalectomy (RLA).

Methods: A retrospective analysis was conducted to include a total of 271 patients diagnosed with PHEO. These patients were separated into two groups: LRA (N=121) and LLA (N=150). The study period spanned from September 2016 to September 2023.

DETAILED DESCRIPTION:
The process of performing an adrenalectomy for pheochromocytoma (PHEO) is difficult due to the significant risk of conversion. The objective of this study was to conduct a comparative analysis of the occurrence and determinants of conversion in left-sided abdominal laparoscopic adrenalectomy (LLA) and right-sided abdominal laparoscopic adrenalectomy (RLA).

Methods: A retrospective analysis was conducted to include a total of 271 patients diagnosed with PHEO. These patients were separated into two groups: LRA (N=121) and LLA (N=150). The study period spanned from September 2016 to September 2023.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral pheochromocytoma of any size, over 18 years old, both males and females

Exclusion Criteria:

* Patients undergoing initial open adrenalectomy, - Additional surgical interventions during total laparoscopic adrenalectomy, - Partial adrenalectomy,

Bilateral PHEOS. Hemorrhagic diathesis, Structural deformity Pregnancy,

- Prior unilateral abdominal surgery, data is absent. The preoperative diagnosis is ambiguous. Hereditary (PHEO), or recurrent PHEO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An analysis of individuals who have undergone TLA and have unilateral PHEO of any size, aged over 18 years, and of both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
conversion | intraoperative
  number of conversion

IPD SHARING:
Plan to Share IPD: No